CLINICAL TRIAL: NCT01748240
Title: Addition of Suberoylanilide Hydroxamic Acid (Vorinostat) to Azacitidine in Patients With Higher Risk Myelodysplastic Syndromes (MDS): a Phase II add-on Study in Patients With Azacitidine Failure.
Brief Title: Addition of Vorinostat to Azacitidine in Higher Risk MDS a Phase II add-on Study in Patients With Azacitidine Failure
Acronym: GFM-AZA-VOR
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: inefficiency
Sponsor: Groupe Francophone des Myelodysplasies (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GFM-Aza-Vor 2012-001401-25
Record Dates: First submitted 2012-12-07; First posted 2012-12-12 (Estimated); Results first posted 2018-08-10 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Azacitidine; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Azacitidine and oral vorinostat (Experimental): Patients who meet eligibility criteria will be administered vorinostat orally at 300mg two times daily for 7 days. AZA will be administered SC at 75 mg/m2/day x 7 consecutive days or at maximum tolerated dose if a dose reduction of AZA was needed before entering the trial with a minimum dose of 50mg/m2/d for 7 consecutive days.
  Each cycle will last 28 days with AZA starting on day 1 of each cycle and vorinostat starting on day 3.
  Interventions: Drug: Azacitidine and oral vorinostat

INTERVENTIONS:
Drug: Azacitidine and oral vorinostat — In patients still responding after six cycles, the drugs will continue to be supplied, and follow up until death or unacceptable tolerance will be continued in all patients.
  Other Names: Suberoylanilide Hydroxamic acid (Vorinostat); Azacitidine (Vidaza)

SUMMARY:
Azacytidine (AZA) is the current standard of care for frontline patient treated with high-risk MDS and is clinically active in all type of MDS, however, 50% of the patients will never respond. Vorinostat is an orally available HDAC inhibitor with clinical activity in MDS and proven in vitro synergy with AZA. Patient treated upfront with a combination of this agents have shown more responses based on phase I/II data. In the present study, we will use the combination of these two drugs to try to create a synergetic effect and generate a response for patients who experienced treatment failure after AZA.

All eligible patients will be treated with Azacitidine and oral vorinostat for 6 cycles of 28 days. Study Design

DETAILED DESCRIPTION:
Patients who meet eligibility criteria will be administered vorinostat orally at 300mg two times daily for 7 days as outlined in table 1.1. AZA will be administered SC at 75 mg/m2/day x 7 consecutive days or at maximum tolerated dose if a dose reduction of AZA was needed before entering the trial with a minimum dose of 50mg/m2/d for 7 consecutive days.

Each cycle will last 28 days with AZA starting on day 1 of each cycle and vorinostat starting on day 3.

Patients will receive 6 cycles unless progression is documented. Patients with a complete remission (CR), partial remission (PR), or hematological improvement (HI), will be treated until progression.

ELIGIBILITY:
Inclusion Criteria:

* Myelodysplastic syndrome (WHO and FAB classified) including: RA, RARS, RCMD, RCMD-RS RAEB , RAEB-t and CMML with WBC < 13000/mm3)
* IPSS score 1.5 or higher (IPSS intermediate-2 and high risk categories) at the beginning of azacitidine,
* Absence of response (CR, PR, marrow CR or HI according to IWG 2006) after a minimum of 6 cycles of azacitidine single agent at 75 mg/m²/d for 7 days per cycle. Patients with a previous dose reduction of AZA may be eligible if the maximum tolerated dose was equal to or above 350mg/m2/cycle (i.e. 50 mg/m²/d for 7 days or 75mg/m2/d for 5 days).
* Age more or egal to 18 years
* ECOG performance status ≤ 2 (cf. appendix 2);
* Patient must have adequate organ function as indicated by the following laboratory values

Renal Serum creatinine or calculated creatinine clearancea < 2 mg/dl OR ≥ 60 mL/min for patients with creatinine levels > 1.5 X institutional ULN Hepatic

Serum total bilirubin ≤ 2.5 X ULN OR direct bilirubin ≤ ULN for patients with total bilirubin levels ≥ 2 mg/dL.

AST (SGOT) and ALT (SGPT) ≤ 2.5 times ULN Alkaline Phosphatase ≤ 5 X ULN If > 2.5 X ULN, then liver fraction should be ≤ 2.5 X ULN a Creatinine clearance should be calculated per institutional standard.

* Patient is known to not be refractory to platelet transfusions.
* Patient ineligible for allogeneic hematopoietic stem cell transplantation at the time of inclusion in the study
* Adherence to the study visit schedule;
* Women of childbearing potential must:

Agree to use effective contraception without interruption throughout the study and for a further 3 months after the end of treatment;

- Men must: Agree to not conceive during the treatment and to use effective contraception during the treatment period (including periods of dose reduction or temporary suspension) and for a further 3 months after the end of treatment if their partner is of childbearing potential.

Agree to learn about the procedures for preservation of sperm.

Exclusion Criteria:

* Patient had prior treatment with an HDAC inhibitor (e.g., depsipeptide or NSC-630176, MS 275, LAQ-824, PXD-101, LBH589, MGCD0103, CRA024781, etc). Patients who have received compounds with HDAC inhibitor-like activity, such as valproic acid, as anti-tumor therapy should not enroll in this study. Patients who have received such compounds for other indications, e.g. valproic acid for epilepsy, may enroll after a 30-day washout period.
* Severe infection or any other uncontrolled severe condition.
* Last dose of AZA was given more than 3 months before entering the trial.
* Patient already enrolled in another therapeutic trial of an investigational drug
* HIV infection or active hepatitis B or C.
* Patient has a known allergy or hypersensitivity to any component of vorinostat or azacitidine.
* Active cancer, or cancer during the year prior to trial entry other than basal cell carcinoma or carcinoma in situ of the cervix or breast.
* Less than 30 days since prior treatment with growth factors (EPO, G-CSF) or non-cytotoxic agents (including low-dose oral chemotherapy); in the event of prior treatment with cytotoxic or demethylating agents, an interval of 3 months is required;
* Patient is on any systemic steroids that have not been stabilized to the equivalent of ≤ 10 mg/day prednisone during the 4 weeks prior to the start of the study drugs.
* Patients with clinical evidence of CNS leukemia.
* Patient has a history of GI surgery or other procedures that might interfere with the absorption or swallowing of the study drugs.
* Women who are or could become pregnant, or who are currently breastfeeding
* Patient eligible for allotransplantation at the time of inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-03; Primary Completion 2013-10 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Prebet, MD, Principal Investigator — Unité d'Hématologie-Institut Paoli Calmettes,Marseille; Pierre Fenaux, MD, Study Director — Hôpital Saint Louis, hematology
Locations (24):
- France (24):
  - CHU d'Angers, Angers
  - CH Annecy, Annecy
  - Hôpital Avignon, Avignon
  - Centre hospitalier de la côte Basque, Bayonne
  - Hôpital Avicenne, Bobigny
  - CHU de Grenoble, Grenoble
  - CH Le mans, Le Mans
  - CH Lyon Sud, Lyon
  - IPC-Unité d'Hématologie 3, Marseille
  - CHU Nantes, Nantes
  - Hôpital Archet1, Nice
  - GHU Caremeau, Nîmes
  - Hôpital Saint Louis, Paris
  - Hopital Saint Louis - AP-HP, Hematology Dpt, Paris
  - Hôpital Saint-Louis, Paris
  - Hopital Cochin-Hematology, Paris
  - Centre Hospitalier Joffre, Perpignan
  - CHU de Haut-Lévèque, Pessac
  - Centre Henri Becquerel, Rouen
  - Hopital Purpan-Medecine interne, Toulouse
  - Hôpital PURPAN, Service d'Hématologie Clinique, Toulouse
  - CHU Bretonneau, Tours
  - CH de Valence, Valence
  - CHU Brabois, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Azacitidine and Oral Vorinostat: Patients who meet eligibility criteria will be administered vorinostat orally at 300mg two times daily for 7 days. AZA will be administered SC at 75 mg/m2/day x 7 consecutive days or at maximum tolerated dose if a dose reduction of AZA was needed before entering the trial with a minimum dose of 50mg/m2/d for 7 consecutive days.
  Each cycle will last 28 days with AZA starting on day 1 of each cycle and vorinostat starting on day 3.
  Azacitidine and oral vorinostat: In patients still responding after six cycles, the drugs will continue to be supplied, and follow up until death or unacceptable tolerance will be continued in all patients.
Period: Overall Study
Arm/Group | Azacitidine and Oral Vorinostat
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Azacitidine and Oral Vorinostat
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 15
Age, Continuous [Median (Full Range); unit: years] | 72 [43 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 15
Region of Enrollment [Number; unit: participants]
  France | 21

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: All eligible patients will be treated with Azacitidine and oral vorinostat for 6 cycles of 28 days.
  The response rate (CR, PR, HI or marrow CR) will be evaluated after six cycles, according to IWG 2006.
  In patients still responding after six cycles, the drugs will continue to be supplied, and follow up until death or unacceptable tolerance will be continued in all patients.
  Complete Response (CR): Bone marrow: less than 5% myeloblasts with Peripheral blood: HI responses).
  Partial remission (RP): Bone marrow blasts decreased by at least 50% but still more than 5% with Peripheral blood: HI responses).
  Marrow CR:Bone marrow: maximum of 5% myeloblasts and decrease by at least 50% over pretreatment
  HI (hematologic improvement)
  * Erythroid response: Hgb increase at least by 1.5 g/dL
  * Platelet response: Increase from less than 20x109/L to more than 20x109/L and by at least 100%
  * Neutrophil response: At least 100% increase and an absolute increase of at least 0.5x109/L
Time Frame: 6 month
Measure: Number (95% Confidence Interval); unit: percentage of response
Arm/Group | Azacitidine and Oral Vorinostat
Number analyzed (Participants) | 21
percentage of response | 5 [0 to 24]

ADVERSE EVENTS:
Arm/Group | Azacitidine and Oral Vorinostat
Serious Adverse Events (participants affected / at risk) | 14/21
Other Adverse Events (participants affected / at risk) | 10/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azacitidine and Oral Vorinostat (N=21)
febrile neutropenia (Blood and lymphatic system disorders) | 14 (14)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azacitidine and Oral Vorinostat (N=21)
diarrhea (Gastrointestinal disorders) | 2 (2) — patients develloping diarrhea
nausea (Gastrointestinal disorders) | 3 (3) — nausea 3/21 (14.28)
vomiting (Gastrointestinal disorders) | 2 (2) — vomiting
constipation (Gastrointestinal disorders) | 2 (2) — cosntipation
undernutrition (Gastrointestinal disorders) | 1 (1) — patients presented the undernutrition

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less